CLINICAL TRIAL: NCT03217279
Title: Typology of Needs and Quality of Life of Stroke Patients and Their Caregivers
Brief Title: Needs Assessment and Quality of Life of Stroke Patients and Their Caregivers
Acronym: TYBRA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0444
Record Dates: First submitted 2017-07-06; First posted 2017-07-14 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Stroke Patients and Their Caregivers
Keywords: stroke-participation; restriction-needs-cohort-patients-caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of Stroke in France is about 150 000 per year. Stroke represents the leading cause of long-term disability. The specificity of stroke is the sequelae polymorphism that can occurs: physical disability, cognitive deficit and sensitive trouble. Then this large extend of sequelae may have a different impact on daily life. Therefore, we have to consider the individual's own resources and in his whole environment to face the situation. We suppose that each situation, each post-stroke disability will have a different social impact in stroke survivors and their caregivers. Nowadays, Barthel Index and Rankin scale are the standards for the assessment of the stroke impact on survivors' daily life. However, what is the real impact of an activity limitation in daily life? How consider the psychosocial impact of stroke only with functional indicators? For this study we will consider handicap and disability in a societal way. In fact, the WHO developed in 2001 the International Classification of functioning, disability and health that allows to bring the concept of participation restriction, this is to say the consequences of a disability in the real life. The ICF allows to bring a conceptual framework of participation restriction.

Psychosocial consequences of stroke are relatively unknown especially in France. According to our hypothesis, patients with major disabilities and their caregivers will experience more psychosocial consequences and participation restriction in terms of emotional health, quality of life and burden. Also, we hypothesize that stroke severity, the typology of disabilities (motor, cognitive and sensorial) will have a different impact on patients and proxys' lifes in terms of psychosocial consequences, participation restriction and quality of life.

TYBRA study is a prospective multicentric cohort study that mixes qualitative and quantitative approaches. The first aim of the quantitative approach is to explore factors related to patients and their caregivers at 6 months that predict participation restriction at 12 months post-stroke. The first aim of the qualitative study is to explore the experience of stroke in minor stroke patients and their proxys.

ELIGIBILITY:
Inclusion Criteria:

* Quantitative study : (patients included in Stroke 69 cohort study)

  * Diagnosis of stroke confirmed by a neurologist or by an emergency doctor after brain imaging (CT or MRI scan)
  * Patients admitted to an emergency department or a neurovascular unit in Rhône department whatever their geographical origin
  * Concerning proxys : Caregivers of patients included in Stroke 69 cohort study and eligible to TYBRA study.

Qualitative study : (patients included in Stroke 69 cohort study)

* Patients included in Stroke 69 cohort study with a diagnosis of stroke confirmed by brain imaging
* Minor stroke (Rankin <1)
* Proxys of minor stroke patients

Exclusion Criteria:

* Patients institutionalized before stroke and/or at 6 months and/or at 12 months
* Patients who have major cognitive trouble
* Stroke during hospitalisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemorrhagic or ischemic stroke patients and their caregivers.
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Change from 6-month participation restriction at 12 months. | At 6 and 12 months post-stroke
  Patients will receive at home questionnaires about the psychosocial consequences of stroke for them and their caregivers at 6 months and 12 months post stroke.
  Scale 2.0 at 12 months. The variable "participation" will be dichotomized in two scores : <50 and >50. A score <50 means that the person presents a significate participation restriction.
Change from 6-month experience of minor stroke for patients and their proxys at 12 months. | Interviews at 6 and 12 months post-stroke
  Semi-structured interviews with stroke patients and their proxys.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No